CLINICAL TRIAL: NCT02538458
Title: Effects of Reduction of the Length of Treatment by Nebulized 3% Hypertonic Saline From 72 to 24 Hours on Clinical Remission, in Children Younger Than 12 Month Hospitalized for Acute Bronchiolitis. BRONDUSAL
Brief Title: Efficacy and Safety of 3% Hypertonic Saline Inhalation (24h vs 72h) to Treat Acute Bronchiolitis in Hospitalized Infants
Acronym: BRONDUSAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-A01335-42
Record Dates: First submitted 2015-08-05; First posted 2015-09-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Bronchiolitis
Keywords: Saline Solution, Hypertonic (3 %); Infant
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Active Comparator): 3 % hypertonic saline up to 72H.
  Interventions: Drug: 3 % hypertonic saline up to 72H
- Placebo control group (Placebo Comparator): * 3 % hypertonic saline up to 24H.
  * Followed by 48 hours of placebo (nebulized 0.9% normal saline).
  Interventions: Drug: 3 % hypertonic saline up to 24H

INTERVENTIONS:
Drug: 3 % hypertonic saline up to 72H — Treatment by inhalation of 3 % hypertonic saline, up to 72H. Test group.
  Other Names: 3 % hypertonic saline
  Arms: Test group
Drug: 3 % hypertonic saline up to 24H — * Treatment by inhalation of 3 % hypertonic saline, up to 24H.
  * followed by 48h of placebo : isotonic saline inhalation. Placebo control group.
  Other Names: palcebo
  Arms: Placebo control group

SUMMARY:
Efficacy/Safety of 3% hypertonic saline inhalation (24H vs 72H) to treat acute bronchiolitis in infants.

DETAILED DESCRIPTION:
In acute bronchiolitis in infants, 3% hypertonic saline nebulizations proved to be efficient, reducing the hospitalization length and clinical severity scores. Among the questions remaining, treatment length is still being discussed in the literature. The trial hypothesis is that the efficiency of a 24 hours treatment by 3% hypertonic saline is not inferior to a 72 hours treatment, in acute bronchiolitis in infants. The primary objective of the study is to compare the efficiency of a 24 hours treatment by 3 % hypertonic saline, versus a 72 hours treatment maximum, on clinical remission, judged by the Wang score measured 72 hours after starting treatment, in children younger than 12 month hospitalized for acute bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* 1st or 2nd episode of acute bronchiolitis, defined by respiratory symptoms episode with initial rhinitis, then cough, then one of the following symptoms : wheezing, crackling, respiratory distress
* Winter epidemic period from November, the 15th, to March the 15th
* Age < 12 months
* Admission Wang score included between 4 and 8
* Infant hospitalized for gravity clinical criteria of severity
* Nebulized 3 % hypertonic saline treatment since less than 24 hours
* Infant with social security card coverage
* Free consent of at least one of the parental authority holder

Exclusion Criteria:

* Pulmonary, cardiac or neurologic chronic underlying disease
* Prematurity < 32 GW
* Asthma (3rd episode or more)
* Admission oxygen saturation level < 85 %, Wang score ≥ 9

Ages: 1 Minute to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Wang score after 72 hours of treatment | 72 hours

SECONDARY OUTCOMES:
Recovery time | From Day 1 to end of the hospitalisation within 2 weeks, assessed at EOS (End of study for the patient, meaning discharge from hospital)
  Secondary outcomes will be assessed during the hospital stay for acute bronchiolitis, from inclusion date until day of hospital discharge, within 2 weeks.
To determine percentage of patient needing transfer to the PICU or use of mechanical ventilation | From Day 1 to end of the hospitalisation, assessed at EOS (End of study for the patient, meaning discharge from hospital)
  Percentage of patient needing transfer to the PICU or use of mechanical ventilation
To assess average time of Oxygen therapy | From Day 1 to end of the hospitalisation, assessed at EOS (End of study for the patient, meaning discharge from hospital)
  average time of Oxygen therapy in days
To assess average time of Tube feeding | From Day 1 to end of the hospitalisation, assessed at EOS (End of study for the patient, meaning discharge from hospital)
  average time of Tube feeding in days.
To determine variation of Wang score during hospitalisation | measured at Day 1, 2, 3, 4 and day of discharge.
  Wang score,
To determine percentage of patient with Adverse Event | From Day 1 to end of the hospitalisation, assessed at EOS (End of study for the patient, meaning discharge from hospital)
  percentage of patient with Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BARBIER, PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Hôpital Couple Enfant, Grenoble, France

REFERENCES:
- [Derived] Beal G, Barbier C, Thoret S, Rubio A, Bonnet M, Mazet R, Ego A, Pin I. Nebulized hypertonic saline 3% for 1 versus 3 days in hospitalized bronchiolitis: a blinded non-inferiority randomized controlled trial. BMC Pediatr. 2019 Nov 8;19(1):417. doi: 10.1186/s12887-019-1804-0. PMID 31699072